CLINICAL TRIAL: NCT03776656
Title: Evaluation of a Treatment With Allopurinol on Autistic Disorders and Epilepsy in Adenylosuccinate Lyase Deficiency (ADSL)
Brief Title: Evaluation of a Treatment With Allopurinol in Adenylosuccinate Lyase Deficiency
Acronym: ADSL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160902J; 2017-002155-28 (EudraCT Number)
Record Dates: First submitted 2018-08-13; First posted 2018-12-17 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Adenylosuccinate Lyase Deficiency
Keywords: Adenylosuccinate lyase; Deficit; Allopurinol; Autism; Epilepsy
MeSH Terms: conditions — Adenylosuccinate lyase deficiency; Autistic Disorder; Epilepsy | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allopurinol (Experimental): Oral administration of Allopurinol (Zyloric®) for 12 months without exceeding 400 mg / day in children and 900 mg / day in adults, with dosage adjustment in case of renal failure
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Daily oral administration
  Other Names: Zyloric®

SUMMARY:
The aim of this study is to evaluate the effectiveness of allopurinol treatment at 12 months on the adaptive and cognitive functioning of patients with adenylosuccinate lyase deficiency (ADSL). The psychiatric evaluation will involve the use of standardized tools prior to initiation of treatment, and will be repeated 6 months and 12 months after the start of treatment.

The decrease in the concentration of SAICAR and S-Ado metabolites, which are markers of adenylosuccinate lyase (ADSL) deficiency, will also be quantified.

Similarly, the efficacy of allopurinol on epileptic seizures for epileptic patients and on electrocardiogram abnormalities will be evaluated secondarily

DETAILED DESCRIPTION:
Adenylosuccinate lyase deficiency (ADSL) is a rare disorder of purine metabolism whose symptoms are mental retardation, autistic disorders, epilepsy, related to the accumulation of succinylpurines: succinylaminoimidazole carboxamide riboside (SAICAr) and succinyladenosine (S- Ado). The S-Ado / SAICAr ratio in the cerebrospinal fluid (CSF) is correlated with the clinical severity: the cerebral toxicity of SAICAr is incriminated. There is no specific treatment.

Based on the work of Gertrude B. Elion (1988 Nobel Prize in Medicine), who reports that allopurinol (a structural analogue of hypoxanthine) can be a substrate for hypoxanthine phosphoribosyltransferase (HPRT) and thus produce allopurinol ribonucleotides with as a first step in the de novo synthesis of purines, investigators tested the hypothesis that treatment with allopurinol in children with ADSL deficiency would reduce the production of the toxic metabolite SAICAr.

This hypothesis was validated in 3 minor patients with biological and clinical improvement.

So the investigators put the phase II, non-comparative study based on 4 visits to Necker-Enfants malades Hospital or La Pitié-Salpêtrière Hospital: Month 0 (before treatment), Month 3, Month 6 and Month 12 after the start of treatment.

After verification of the inclusion criteria and information of the parents or the patient or guardian, signature of the consent and inclusion of the patient:

* Clinical and neurological evaluation;
* Psychiatric assessment with standardized tests;
* Biological evaluation: determination of urinary and plasma metabolites (SAICAr, S-Ado, ...) Experimental treatment: Allopurinol (Zyloric®) will be administered orally for 12 months without exceeding 400 mg / day in children and 900 mg / day in adults, with dosage adjustment in case of renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Child (minimum age 18 months) or adult with adenylosuccinate lyase; deficiency (ADSL) confirmed by quantification of SAICAr and S-Ado urinary;
* Girls / women of childbearing age must:

  * have a negative pregnancy test;
  * agree to use a reliable method of contraception from the baseline visit to the last dose of study treatment
* Consent of the patient, his parents or his legal representative;
* Beneficiary of social security (affiliated or entitled).

Exclusion Criteria:

* Refusal of the child, his parents or the patient or his representative;
* Allergy known to allopurinol or to one of the constituents of the product (lactose in particular);
* Patients treated with Antipurines (azathioprine, mercaptopurine);
* Patients treated with vidarabine, cytotoxic drugs (eg cyclophosphamide, doxorubicin, bleomycin, procarbazine, alkyl halides), ciclosporin, or didanosine
* Renal failure characterized by creatinine clearance <80 ml/mn
* Hepatic insufficiency
* Medullary insufficiency but possibly serious
* Breastfeeding
* Pregnancy or wishing to conceive during the study period

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Measurement of adaptive functional improvement : composite total score for Vineland II adaptive behaviour Scale | 12 months
  to assess Efficacy of Allopurinol (Zyloric)® treatment from Baseline : For each scale : Mean : 100 SD : 15
  * Adaptive behaviour composite : Range 20 to 180 -Domains scores : Range 20 to 140 -Communication : Range 20 to 140 -Daily living skills : Range 20 to 140 -Socialization : 20 to 140 -Motor skills : 20 to 140 For each scale values are considered to be better or worse outcome :High 130 to 140 -Moderately High 115 to 129 -Adequate 86 to 114 -Moderately Low 71 to 85 -Low 20 to 70 Total score is obtained by summing the subdomains scores

SECONDARY OUTCOMES:
Evolution of the Scores of different subdomains Vineland II scale from baseline | at 0, 6 months and 12 months
  Clinical evolution for developmental and cognitive assessment
Evolution of the Psycho-Educative Profile (PEP III/R) from baseline | at 0, 12 months
  Clinical evolution for developmental and cognitive assessment
Evolution of the Score ADI-R (Autism Diagnostic Interview-Revised) from baseline | at 0, 12 months
  Clinical evaluation for autistic symptoms : scale ranges :
  * A : Social interactions: 0 to 30 (significative if >10)
  * B : Communication : 0 to 26 (significative if > 7 or 8)
  * C : Repetitive and restricted interests : 0 to 16 (significative if >3)
  * D : Developmental abnormality present before 36 months : 0 to 5 (significative if >1)
  better score : 0 (non autistic) - worse score : the higher score is the worst
Evolution of the Score ADOS-2 (Autism Diagnostic Observation Schedule 2) from baseline | at 0, 12 months
  Clinical evaluation for autistic symptoms. Scale ranges :
  * A : Socialization : social interactions and communication : 0 to 20 (social interactions : 0 to 6 -communication : 0 to 14)
  * B : Restricted and repetitive interests : 0 to 8
  * Total : A+B : 0 to 28
  Autism : total score>12 - Autism Spectrum Disorder : total score >8
  Better score : 0 - Worse score : the highest score is the worst
Evolution of the Score on Conners hyperactivity Scale | at 0, 6 months and 12 months
  Clinical evolution for behavioral disorders and adaptive functioning
  Conners Scale for Parents :
  - Subscales : Behavioural difficulties (items 2-8-14-19-20-27-35-39) : 0 to 24 Learning difficulties (items 10-25-31-37) : 0 to 12 Somatisation (items 32-41-43-44) : 0 to 12 Impulsivity, hyperactivity (items 4-5-11-13): 0 to 12 Anxiety (items 12-16-24-47): 0 to 12
  -Hyperactivity index : sum of the items (4-7-11-13-14-25-31-33-37-38) divided by 10 : 0 to 3
  Conners Scale for teachers :
  - Subscales : Behavioural difficulties (items 4-5-6-10-11-12-23-27) : 0 to 24 Impulsivity, hyperactivity (items 1-2-3-8-14-15-16) : 0 to 21 Inattention, passivity (items 7-9-18-20-21-22-26-28) : 0 to 24
  -Hyperactivity index (sum of the items 1-5-7-8-10-11-14-15-21-26 divided by 10) : 0 to 3
  Better score : 0 - Worse score : the highest score is the worst -Hyperactivity index : Significative if> 1,5
Evolution of the Score on ABC scale (Aberrant Behaviour Checklist) | at 0, 6 months and 12 months
  Clinical evolution for behavioral disorders and adaptive functioning scale ranges :
  * Irritability : 0 to 45
  * Lethargy : 0 to 48
  * Stereotypy : 0 to 21
  * Hyperactivity : 0 to 48
  * Inappropriate speech : 0 to 12
  Better score : 0 -Worse score : the highest score is the worst on each scale- there is no total score
Evolution of SAICAr levels in the urine | at 0, 6 months and 12 months
  Evolution of the quantity of urinary metabolites from Baseline
Evolution of S-Ado levels in the urine | at 0, 6 months and 12 months
  Evolution of the quantity of urinary metabolites from Baseline
Evolution of SAICAr levels in the blood | at 0, 6 months and 12 months
  Evolution of the quantity of plasma metabolites from Baseline
Evolution of S-Ado levels in the blood | at 0, 6 months and 12 months
  Evolution of the quantity of plasma metabolites from Baseline
Evolution of the number of seizures from Baseline for epileptic patients | at 0 and 12 months
  at baseline, performing neurological examinations and interrogation
Evolution of antiepileptic treatments from Baseline for epileptic patients | at 0 and 12 months
  at baseline, performing neurological examinations and interrogation
Evolution of electroencephalogram tracing from Baseline for epileptic patients | at 0 and 12 months
  normal/abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Pascale De LONLAY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Irène CEBALLOS-PICOT, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Laurence ROBEL-GALLI, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - LA PITIE-SALPETRIERE Hospital, AP-HP, Paris
  - Department of Pediatry. Reference centre of Hereditary diseases of the metabolism of child and adult. Necker - Enfants malades Hospital, Paris

IPD SHARING:
Plan to Share IPD: No